CLINICAL TRIAL: NCT05025605
Title: A Randomized, Double-blind, Placebo-controlled Study to Determine Efficacy and Safety of BXCL501 in Agitation Associated With Pediatric Schizophrenia and Bipolar Disorder
Brief Title: Determining Efficacy and Safety of BXCL501 in Agitation Associated With Pediatric Schizophrenia and Bipolar Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioXcel Therapeutics Inc (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BXCL501-105
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia; Schizo-Affective Disorder; Schizophreniform; Schizophrenic; Bipolar Disorder I; Bipolar Disorder II
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Study will randomize subjects in Group one 1:1:1 to receive BXCL501 80 μg, BXCL501 120 μg, or matching placebo film; Group two 2:1 to receive BXCL501 60 μg or matching placebo film
Who Masked: Participant, Investigator
Masking Description: Double-Blind, Placebo-controlled
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 80 Micrograms (Experimental): Sublingual film containing 80 micrograms Dexmedetomidine
  Interventions: Drug: BXCL501 80 Micrograms
- 120 Micrograms (Experimental): Sublingual film containing 120 micrograms Dexmedetomidine
  Interventions: Drug: BXCL501 120 Micrograms
- Placebo (Placebo Comparator): Sublingual Placebo film
  Interventions: Drug: Placebo Film
- 60 Micrograms (Experimental): Sublingual film containing 60 micrograms Dexmedetomidine Europe Only
  Interventions: Drug: BXCL501 60 Micrograms

INTERVENTIONS:
Drug: BXCL501 80 Micrograms — Sublingual film containing 80 Micrograms BXCL501
  Other Names: Dexmedetomidine
  Arms: 80 Micrograms
Drug: Placebo Film — Matching Sublingual Placebo film
  Other Names: Placebo
  Arms: Placebo
Drug: BXCL501 120 Micrograms — Sublingual film containing 120 Micrograms BXCL501
  Other Names: Dexmedetomidine
  Arms: 120 Micrograms
Drug: BXCL501 60 Micrograms — Sublingual film containing 60 Micrograms BXCL501 Europe Only
  Other Names: Dexmedetomidine
  Arms: 60 Micrograms

SUMMARY:
This is a study of the efficacy and safety of BXCL501 in children and adolescents with acute agitation and either bipolar disorder or schizophrenia.

DETAILED DESCRIPTION:
The study will enroll approximately 140 subjects randomized to dose regimens of 80 µg or 120 µg BCXL501 or placebo (Group one), or 60 µg BCXL501 or placebo (Group two; Europe only). Subjects with acute agitation will include male and female children and adolescents who are either newly admitted to a hospital setting or already admitted and experiencing acute agitation. Subjects will be domiciled in a clinical research setting or hospitalized to remain under medical supervision while undergoing screening procedures to assess eligibility. Efficacy and safety assessments will be conducted periodically before and after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 10-17 years, inclusive, with bipolar disorder (DSM-5 criteria) and 13-17 years, inclusive, in subjects with schizophrenia (DSM-5 criteria).
2. Patients who are judged to be clinically agitated at Screening and Baseline with a total score of ≥14 on the 5 items comprising the PANSS Excited Component (PEC).
3. Patients who have a score of ≥ 4 on at least 1 of the 5 items on the PEC at Baseline.
4. Participants who agree to use a medically acceptable and effective birth control method

Exclusion Criteria:

1. Patients with agitation caused by acute intoxication, including alcohol or drugs of abuse (with the exception of THC) during urine screening.
2. Use of benzodiazepines or other hypnotics or oral or short-acting intramuscular antipsychotic drugs in the 4 hours before study treatment.
3. Patients who are judged to be at significant risk of suicide.
4. Patients with serious or unstable medical illnesses.
5. Patients who have received an investigational drug within 30 days prior to the current agitation episode.
6. Patients who are considered by the investigator, for any reason, to be an unsuitable candidate for receiving the study drug.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in the Positive and Negative Syndrome Scale - Excited Component (PEC) total score | 120 minutes - Group one only
  The Positive and Negative Syndrome Scale - Excited Component (PEC) comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored 1 (minimum) to 7 (maximum). The PEC, the sum of these 5 subscales, thus ranges from 5 (absence of agitation) to 35 (extremely severe)

SECONDARY OUTCOMES:
Absolute change from baseline in the Positive and Negative Syndrome Scale - Excited Component (PEC) total score | 90, 60, 45, 30, 20,10 minutes - Group one only
  The Positive and Negative Syndrome Scale - Excited Component (PEC) comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored 1 (minimum) to 7 (maximum). The PEC, the sum of these 5 subscales, thus ranges from 5 (absence of agitation) to 35 (extremely severe)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Risinger, MD, Study Chair — BioXcel Therapeutics
Locations (5):
- United States (5):
  - BioXcel Clinical Research Site, Anaheim, California
  - Bioxcel Clinical Research Site, Hialeah, Florida
  - BioXcel Clinical Research Site, Atlanta, Georgia
  - Bioxcel Clinical Research Site, Decatur, Georgia
  - BioXcel Clinical Research Site, DeSoto, Texas